CLINICAL TRIAL: NCT01381861
Title: A Phase 2 Evaluation of TRC105 in the Treatment of Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: Evaluation of TRC105 in the Treatment of Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105OC201
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Recurrent Ovarian Cancer; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carotuximab (TRC105) alone (Experimental): Single arm, open label Carotuximab (TRC105) alone therapy dosed at 10 mg/kg administered intravenously over 1 to 4 hours on days 1, 8, 15 and 22 of each 28 day cycle
  Interventions: Biological: Carotuximab (TRC105)

INTERVENTIONS:
Biological: Carotuximab (TRC105) — Carotuximab (TRC105) 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
  Other Names: TRC105; NSC#754227

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TRC105 in patients with recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.

DETAILED DESCRIPTION:
Angiogenesis plays a central role in the progression of epithelial ovarian cancer. In mouse models, VEGF-inhibitors diminish ovarian tumor growth, metastasis and malignant ascites formation. Independent Phase 2 trials have demonstrated single-agent activity for bevacizumab in recurrent ovarian cancer, and randomized controlled Phase 3 trials are ongoing in the first-line setting (GOG 0218 and ICON-7) and for recurrent disease (GOG 0213, OCEANS).

TRC105 is an antibody to CD105, an important non-VEGF angiogenic target on vascular endothelial cells. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models. In a Phase 1 study of advanced solid tumors, TRC105 therapy caused a global reduction in angiogenic biomarkers and reduced tumor burden at doses that were well-tolerated. We hypothesize that TRC105 will have single-agent activity in recurrent ovarian cancer. By targeting a non-VEGF pathway, TRC105 has the potential to complement VEGF inhibitors which could represent a major advance in ovarian cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma
* Measurable disease per RECIST 1.1
* At least one "target lesion" per RECIST 1.1
* Patients must have GOG Performance Status of 0 or 1
* Patients must have a life expectancy of ≥ 3 months
* Resolution of all acute toxic effects of prior therapy
* Free of active infection requiring antibiotics
* Must have had one prior platinum-based chemotherapeutic regimen for management of primary disease
* Patients could have received one additional cytotoxic regimen for management of recurrent disease
* Prior therapy directed at the malignant tumor, including hormonal and immunologic agents, must be discontinued at least three weeks prior to registration. Continuation of hormone replacement therapy is permitted.
* Adequate bone marrow function, renal function, hepatic function, neurologic function, blood coagulation parameters
* Negative serum pregnancy test and effective form of contraception for patients of childbearing potential

Exclusion Criteria:

* Previous treatment with TRC105
* Current treatment on another therapeutic clinical trial
* Receipt of an investigational agent within 28 days of starting study treatment
* Serious, non-healing wounds, ulcers, or bone fractures.
* Active bleeding or pathologic conditions that carry a high risk of bleeding
* Patients with tumor involving major vessels or transmural bowel wall involvement by tumor
* Use of thrombolytic or anticoagulant agents (except heparin to maintain i.v. catheters) within 10 days prior to the first dose of TRC105
* History of deep venous thrombosis (DVT)(except patients who have received adequate anticoagulation are eligible, and may continue on anticoagulation if appropriate)
* History of peptic ulcer disease or erosive gastritis within the past 6 months
* Known active viral or nonviral hepatitis
* History or evidence of CNS disease
* Clinically significant cardiovascular disease
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human, chimeric, or humanized antibodies
* Pregnant or nursing
* Under the age of 18
* Patients with or with anticipation of invasive procedures including major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to treatment with TRC105
* History of other invasive malignancies, except non-melanoma skin cancer and other cancers that have been treated with no evidence of disease within the last 3 years
* History of primary endometrial cancer diagnosed within the last 5 years, unless all of the following conditions are met: Stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO Grade 3 lesions
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last five years are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed > 3 years prior to registration, and patient remains free of recurrent or metastatic disease
* Prior radiotherapy to any portion of the abdominal cavity or pelvis
* Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Theuer, MD, Study Director — TRACON Pharmaceuticals
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Indiana University-Bren and Melvin Simon Cancer Center, Indianapolis, Indiana
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and enrolled at 7 US sites
Groups:
- TRC105: Chimeric monoclonal antibody (TRC105) to CD105: 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
Period: Overall Study
Arm/Group | TRC105
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Total number of patients enrolled in the trial who received at least a portion of a dose of TRC105. Screen-failure patients are not included in the overall baseline analysis population.
Arm/Group | TRC105
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: Years] | 59.8 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate After 6 Months of Treatment on Study
Description: Number of patients ongoing within the study who have not progressed after 6 months of treatment
Time Frame: 6 months
Population: This population will include all patients enrolled in the study who receive at least 1 dose of TRC105 study medication and who undergo at least one on study efficacy assessment or expire due to progressive disease prior to the first efficacy assessment.
Measure: Number; unit: participants
Arm/Group | TRC105
Number analyzed (Participants) | 23
participants | 0

2. Primary Outcome: Proportion of Patients Who Have Objective Tumor Response
Description: Proportion of patients who have objective tumor response (complete or partial) by RECIST 1.1
Time Frame: Every 2 cycles
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TRC105
Number analyzed (Participants) | 22
participants | 0

3. Primary Outcome: Adverse Events
Description: Frequency of adverse events as assessed by NCI CTCAE (Version 4.0)
Time Frame: 28 days
Population: All patients who received at least a portion of a dose of TRC105.
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105
Number analyzed (Participants) | 23
Participants
  Anemia (Grade 3 Suspected Reaction) | 4
  Fatigue (Grade 3 Suspected Reaction) | 1
  Headache (Grade 3 Suspected Reaction) | 2
  Migraine (Grade 3 Suspected Reaction) | 1
  Epistaxis (Grade 3 Suspected Reaction) | 1

4. Secondary Outcome: CA-125 Response Rate
Description: CA-125 response rate by GCIG criteria
Time Frame: Every 2 cycles
Population: All patients who received at least a portion of a dose of TRC105
Measure: Number; unit: participants
Arm/Group | TRC105
Number analyzed (Participants) | 23
participants
  CA-125 Decrease | 7
  CA-125 Increase | 16

5. Secondary Outcome: Serum Concentrations of TRC105
Description: Median peak and trough concentration of TRC105 by ELISA in ug/mL
Time Frame: Cycle 1 Day 15
Population: All patients who received at least a portion of a TRC105 dose
Measure: Median (Full Range); unit: ug/mL
Arm/Group | TRC105
Number analyzed (Participants) | 23
ug/mL
  Median Trough Concentration Cycle 1 Day 15 | 47.4 [0 to 93.1]
  Median Peak Concentration Cycle 1 Day 15 | 274.5 [114 to 425]

6. Secondary Outcome: TRC105 Immunogenicity
Description: TRC105 Anti-Drug Antibody (ADA) Immunogenicity by ELISA
Time Frame: 1 year
Population: All patients that received at least a portion of TRC105
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105
Number analyzed (Participants) | 17
Participants
  Patients with Positive Treatment Emergent ADA | 7
  Patients with Negative Treatment Emergent ADA | 10

7. Secondary Outcome: Severity of Adverse Events
Description: Severity of adverse events by NCI CTCAE
Time Frame: 28 days post last dose of TRC105
Population: All patients who received at least a portion of a dose of TRC105.
Measure: Number; unit: participants
Arm/Group | TRC105
Number analyzed (Participants) | 23
participants
  Serious Adverse Events | 6
  TRC105 Related Serious Adverse Events | 1
  No Serious Adverse Events | 16

8. Secondary Outcome: Overall Survival
Description: Median overall survival
Time Frame: 2 years
Population: Data not collected
Arm/Group | TRC105
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for at least 28 days after the last dose of TRC105 study drug for adverse events, on average approximately 4 months.
Arm/Group | TRC105
All-Cause Mortality (participants affected / at risk) | 3/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 (N=23)
Headache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Disease progression (General disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 (N=23)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 9 (9)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Gingival pain (Gastrointestinal disorders) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 2 (2)
Disease progression (General disorders) | 3 (3)
Fatigue (General disorders) | 12 (12)
Mucosal inflammation (General disorders) | 3 (3)
Pyrexia (General disorders) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 13 (13)
Migraine (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Epistaxis (Vascular disorders) | 17 (17)
Flushing (Vascular disorders) | 6 (6)
Gingival bleeding (Vascular disorders) | 11 (11)
Hot flush (Vascular disorders) | 2 (2)
Telangiectasia (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less